CLINICAL TRIAL: NCT06175910
Title: Safety and Efficacy of Percutaneous Nephrolithotripsy Versus Retrograde Intrarenal Surgery for Obese Patients With Pelvic 1.5:3 cm Renal Stones
Brief Title: Postoperative Outcomes of PCNL vs RIRS in Obese Patients With Pelvic 1.5:3 cm Renal Stones
Acronym: PCNL VS RIRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: bassem metwally (Other)
Collaborators: Helwan University (Other)
Responsible Party: Sponsor-Investigator, bassem metwally, Principal Investigator, Helwan University
Organization: Helwan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 72 - 2020
Record Dates: First submitted 2023-11-21; First posted 2023-12-19 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Renal Stones
Keywords: Renal Stones; Retrograde Intrarenal Surgery (RIRS); Percutaneous Nephrolithotomy (PCNL); Stone-free Rate; Obese Patients
MeSH Terms: conditions — Nephrolithiasis | interventions — Nephrolithotomy, Percutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- percutaneous nephrolithotomy (Active Comparator): 60 patients were undergone percutaneous nephrolithotomy, three patients were lost in follow up and one case was excluded due to stricture urethra. So, the investigators analysed 56 patients
  Interventions: Procedure: percutaneous nephrolithotomy
- retrograde intrarenal surgery (Active Comparator): 60 patients were undergone retrograde intrarenal surgery, one patient was lost in follow up and one case was aborted due to narrow ureter & DJ was applied. So, the investigators analysed 58 patients.
  Interventions: Procedure: retrograde intrarenal surgery

INTERVENTIONS:
Procedure: percutaneous nephrolithotomy — A 7 Fr ureteric catheter was placed into the ipsilateral ureteric orifice. The patients were then placed in the prone position. Opacification of the pelvicalyceal system was performed. The puncture was done by a 22-guage puncture needle was advanced into the posterior lower calyx under fluoroscopic guidance. After successful access is established, a 0.035-inch curved guide wire was advanced through the puncture needle into the kidney. The central Alkane Rod was passed over the guide wire. Under fluoroscopic guidance serial Amplatz dilators up to 30 Fr were advanced over central Alkane rod and guide wire. Then 30 Fr long Amplatz sheath was advanced over the last dilator.
  26 Fr rigid long nephroscope used for stone fragmentation and retrieval. Stone fragmentation was done by pneumatic Swiss Lithoclast. Fragments removal was done using toothed peanut stone retrieval forceps.
  Other Names: flexible ureteroscope
  Arms: percutaneous nephrolithotomy
Procedure: retrograde intrarenal surgery — urethrocystoscopy was carried out then inserting of a 7F open ended ureteral catheter over the 0.035-inch straight floppy tip guide wire in the working channel of the 22Fr cystoscope under fluoroscopic guidance, access to the ureter was made.
  Teflon ureteric dilators are used to dilate the distal ureter till 14 FR. ureteral access sheath placement 12 or 14 Fr. OTU, a disposable digital flexible ureteroscope, is then used then the tip of a 272 m holmium laser fiber is placed on the surface of the stone for fragmentation.
  Intra renal lithotripsy was carried out using a 30 W Holmium: YAG laser (Sphinx Jr.) via a 272 m silica quartz laser fiber. 1.9 Fr tipless nitinol baskets were finally used to remove the large fragments. A Double-J (6 Fr) stent is generally applied at the end of the procedure, and a urethral catheter was applied.
  Other Names: flexible ureteroscope
  Arms: retrograde intrarenal surgery

SUMMARY:
This prospective randomized comparative study was done at Helwan University Hospital. It was conducted on 120 patients with unilateral pelvic renal stones from 1.5 to 3 cm in largest diameter who was admitted through duration to compare the two procedures differences in terms of complications, analgesic use, hospital stay, operational time, and stone-free rates.

DETAILED DESCRIPTION:
In this study, 182 patients were assessed for eligibility; 62 patients were excluded, 48 of which were not meeting our inclusion criteria and 14 patients declined to participate in the study as detailed in the CONSORT flowchart

After meeting our inclusion and exclusion criteria, 120 patients were thoroughly informed about the study and after feeling well about participating in it a written informed consent was taken from them. Patients were randomly divided into two equal groups using a closed envelope technique into:

* Group A: 60 patients were undergone percutaneous nephrolithotomy, three patients were lost in follow up and one case was excluded due to stricture urethra. So, the investigators analysed 56 patients.
* Group B: 60 patients were undergone retrograde intrarenal surgery, one patient was lost in follow up and one case was aborted due to narrow ureter & DJ was applied. So, the investigators analysed 58 patients

All participants were submitted to preoperative assessment:

History-taking, clinical examination, laboratory examination (urine analysis, urine culture and sensitivity, blood urea, creatinine levels, complete blood counts, and coagulation profile), Imaging modalities: ultrasonography, plain radiograph of kidney-ureter-bladder (KUB) and non-contrast computed tomography (CT).

The following data were recorded:

The information on the patient's characteristics (age and gender), the characteristics of the kidney stones (size and laterality), the length of the procedure in minutes from the induction of anesthesia till the end of procedure (insertion of the nephrostomy in PCNL and the insertion of the urethral catheter in RIRS), and intraoperative complications with a focus on bleeding, stone migration, and extravasation.

Postoperative data and follow up:

1. Stone clearance: The patients had radiographic evaluation during the first- and fourth-weeks following surgery, using spiral CT without contrast for radiolucent stones and simple KUB for stones that were radiopaque.

   Stone-free or stone residual < 3 mm after just one session of the therapy were considered successful outcomes.
2. Postoperative fever < 38 degrees.
3. Postoperative bleeding.
4. Hospital stay from the day of operation till the day of discharge (in days).
5. The need for analgesics.

ELIGIBILITY:
Inclusion Criteria:

* Obese adult patients with body mass index ≥30
* aged ≥ 18 years
* unilateral pelvic renal stone from 1.5 to 3 cm in largest diameter.

Exclusion criteria:

* A single kidney
* renal impairment (serum creatinine > 1.4 mg/dl)
* patients with uncontrolled co-morbidities (hypertension, diabetes mellitus, cardiac disease, chest disease)
* active Urinary tract infection
* ureteric or bladder stones
* anatomic renal abnormalities (congenital renal malformations such as horseshoe kidney, polycystic kidney disease, etc.)
* people with severe skeletal deformity
* pregnant women
* history of ureteric strictures
* uncorrectable bleeding disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
stone free rate | one month
  Stone-free or stone residual < 3 mm after just one session of the therapy were considered successful outcomes.Data were gathered, edited, coded, and entered into IBM SPSS version 23 of the Statistical Package for Social Science.

SECONDARY OUTCOMES:
complications | two weeks
  fever >38 ,intra or postoperative bleeding, Pelvicalyceal system injury.Data were gathered, edited, coded, and entered into IBM SPSS version 23 of the Statistical Package for Social Science.
operation time | during procedure ( till five hours)
  the length of the procedure in minutes from the induction of anesthesia till the end of procedure .Data were gathered, edited, coded, and entered into IBM SPSS version 23 of the Statistical Package for Social Science.
hospital stay | from the day of procedure till the day of discharge from hospital (two weeks)
  from the day of operation till the day of discharge (in days).Data were gathered, edited, coded, and entered into IBM SPSS version 23 of the Statistical Package for Social Science.
analgesic use | from the day of procedure till the day of discharge from hospital (two weeks)
  Number of patients need analgesic in form of non steroidal anti inflammatory drugs. Data were gathered, edited, coded, and entered into IBM SPSS version 23 of the Statistical Package for Social Science.

CONTACTS AND LOCATIONS:
Overall Officials: bassem A metwally, master, Principal Investigator — Helwan University
Locations (1):
- Helwan University, Cairo, Helwan, Egypt